CLINICAL TRIAL: NCT05454917
Title: Evaluation of Intraoperative V/Q Mismatch and Compliance Trajectories as Predictors of Pulmonary Postoperative Complications in Patients Undergoing Major Surgery
Brief Title: Evaluation of V/Q Mismatch as Predictor of Pulmonary Postoperative Complications in Patients Undergoing Major Surgery
Acronym: VQppc
Status: Completed | Type: Observational
Sponsor: Università degli Studi di Ferrara (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Principal Investigator, Savino Spadaro, Principal Investigator, Università degli Studi di Ferrara
Other Study IDs: VQppc
Record Dates: First submitted 2022-07-04; First posted 2022-07-12 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Anesthesia; Postoperative Complications; Mechanical Ventilation Complication
Keywords: Anesthesia; Pulmonary postoperative complications; ALPE; Ventilation/perfusion mismatch
MeSH Terms: conditions — Postoperative Complications; Respiratory Aspiration | interventions — Perfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing surgery: Mechanical measures, VQ mismatch evaluation
  Interventions: Device: Measure of ventilation/perfusion (V/Q) mismatch using Beacon ALPE (Automatic Lung Paramether Estimator)

INTERVENTIONS:
Device: Measure of ventilation/perfusion (V/Q) mismatch using Beacon ALPE (Automatic Lung Paramether Estimator) — Evaluation of intraoperative V/Q mismatch using the Beacon ALPE during anesthesia.

SUMMARY:
Pulmonary postoperative complications (PPC) are among the main causes of surgical complications affecting both postoperative morbidity and mortality. Little is known about the effect of intraoperative VQ mismatch on the occurrence of PPC. In this trial the investigators will evaluate if intraoperative VQ mismatch may predict PPC in a population of patients undergoing major surgery.

DETAILED DESCRIPTION:
Pulmonary postoperative complications (PPC) are among the main causes of surgical complications affecting both postoperative morbidity and mortality. Little is known about the effect of intraoperative VQ mismatch on the occurrence of PPC.

PPC are classically considered associated to the occurrence of intraoperative atelectasis, and therefore to the development of a certain amount of shunt, but this concept have been recently questioned.

Recent studies showed indeed that, despite age is one of the main determinants of PPCs, increasing age is not associated to the increase of intraoperative shunt. Shunt therefore may not be the main determinant of PPC.

In this trial the investigators will evaluate if other causes of intraoperative VQ mismatch (e.g. low V/Q, high V/Q, dead space) may predict PPC in a population of patients undergoing major surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-90 years
* Major elective surgery with general anesthesia
* Intraoperative cannulation of the radial artery for invasive pressure monitoring

Exclusion Criteria:

* Thoracic surgery with one lung ventilation
* Refuse to participate
* Emergency surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing general anesthesia for elective major surgery (non-thoracic).
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Occurrence of Pulmonary postoperative complications | In the first 7 days after surgery
  Definition derived from the ESA-ESICM joined taskforce on perioperative outcome measures.

SECONDARY OUTCOMES:
Intraoperative mechanical measures (pressures) | During surgery
  Intraoperative evaluation of:
  * Peak pressure (Ppeak), cmH2O
  * Plateau pressure (Pplat), cmH2O
  * Total PEEP (PEEP total), cmH2O
Intraoperative drug administration | During surgery
  Evalation of anesthetic drugs administered during surgery by the treating physician.
Intraoperative arterial pressure | During surgery
  Evaluation during surgery of:
  * systolic pressure (mmHg)
  * diastolic pressure (mmHg)
Intraoperative heart rate | During surgery
  evaluation of
  - Heart rate (beats/min)
V/Q mismatch | During anesthesia
  Evaluation of V/Q mismatch
fluid balance | During surgery
  Evaluation of patients fluid intake and fluid balance during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Savino Spadaro, MD, PhD, Study Director — Università degli Studi di Ferrara; Gaetano Scaramuzzo, MD, Principal Investigator — Università degli Studi di Ferrara
Locations (1):
- Azienda Ospedaliero Universitaria Sant'Anna, Ferrara, Italy

REFERENCES:
- [Background] Hedenstierna G, Tokics L, Scaramuzzo G, Rothen HU, Edmark L, Ohrvik J. Oxygenation Impairment during Anesthesia: Influence of Age and Body Weight. Anesthesiology. 2019 Jul;131(1):46-57. doi: 10.1097/ALN.0000000000002693. PMID 31045901
- [Background] Miskovic A, Lumb AB. Postoperative pulmonary complications. Br J Anaesth. 2017 Mar 1;118(3):317-334. doi: 10.1093/bja/aex002. PMID 28186222
- [Background] Spadaro S, Grasso S, Karbing DS, Santoro G, Cavallesco G, Maniscalco P, Murgolo F, Di Mussi R, Ragazzi R, Rees SE, Volta CA, Fogagnolo A. Physiological effects of two driving pressure-based methods to set positive end-expiratory pressure during one lung ventilation. J Clin Monit Comput. 2021 Oct;35(5):1149-1157. doi: 10.1007/s10877-020-00582-z. Epub 2020 Aug 20. PMID 32816177
- [Background] Jammer I, Wickboldt N, Sander M, Smith A, Schultz MJ, Pelosi P, Leva B, Rhodes A, Hoeft A, Walder B, Chew MS, Pearse RM; European Society of Anaesthesiology (ESA) and the European Society of Intensive Care Medicine (ESICM); European Society of Anaesthesiology; European Society of Intensive Care Medicine. Standards for definitions and use of outcome measures for clinical effectiveness research in perioperative medicine: European Perioperative Clinical Outcome (EPCO) definitions: a statement from the ESA-ESICM joint taskforce on perioperative outcome measures. Eur J Anaesthesiol. 2015 Feb;32(2):88-105. doi: 10.1097/EJA.0000000000000118. PMID 25058504